CLINICAL TRIAL: NCT00579345
Title: A Phase III, Single-Blind, Multi-Center, Extension Study to Evaluate Safety and Tolerability of a Trivalent Subunit Influenza Vaccine Produced Either in Mammalian Cell Culture or in Embryonated Hen Eggs in Adult and Elderly Subjects Who Participated in Study V58P4, With Subset Analyses of Immunogenicity and Evaluation of Concomitant Polysaccharide Pneumococcal Vaccine (Elderly).
Brief Title: Second Extension Study to Evaluate Safety and Tolerability of Influenza Vaccines in Adults and Elderly, and to Evaluate Immunogenicity and Concomitant Vaccination With Pneumococcal Vaccine in a Subgroup
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V58P4E2; 2006-003077-27
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Results first posted 2011-10-10 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2012-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- cTIV (Experimental): Cell culture derived seasonal trivalent influenza vaccine (cTIV)
  Interventions: Biological: Cell culture derived seasonal trivalent influenza vaccine (cTIV)
- eTIV_a (Active Comparator): Influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a)
  Interventions: Biological: Influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a).
- FLU (cTIV or eTIV_a) (Experimental): Cell culture derived seasonal trivalent influenza vaccine (cTIV) or influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a).
  Interventions: Biological: cTIV or eTIV_a
- FLU (cTIV or eTIV_a) + PV (Active Comparator): 23-valent Pneumococcal vaccine (PV) concomitantly administered with cell culture derived seasonal trivalent influenza vaccine (cTIV) or influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a).
  Interventions: Biological: cTIV+PV OR eTIV_a+PV

INTERVENTIONS:
Biological: Cell culture derived seasonal trivalent influenza vaccine (cTIV) — cell cultured trivalent influenza vaccine (cTIV) vaccine administered as 0.5 mL single dose in the deltoid muscle, preferably of the non-dominant arm.
  Arms: cTIV
Biological: Influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a). — egg based trivalent influenza vaccine (eTIV_a) administered as 0.5 mL single dose in the deltoid muscle, preferably of the non-dominant arm.
  Arms: eTIV_a
Biological: cTIV or eTIV_a — 0.5 mL, Single dose of either cell cultured trivalent influenza vaccine (cTIV) or egg based trivalent influenza vaccine eTIV_a administered.
  Arms: FLU (cTIV or eTIV_a)
Biological: cTIV+PV OR eTIV_a+PV — 0.5 mL, Single dose of either cell culture derived seasonal trivalent influenza vaccine (cTIV) or influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a) administered concomitantly with 23-valent pneumococcal polysaccharide vaccine (PV).
  Arms: FLU (cTIV or eTIV_a) + PV

SUMMARY:
The study primarily aims to evaluate immunogenicity and safety of influenza vaccines (cell culture derived seasonal trivalent influenza vaccine (cTIV) or influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a)) when administered alone and when administered concomitantly with pneumococcal polysaccharide vaccine (PV) in elderly subjects. The study also aimed to evaluate safety and immunogenicity (subset) of annual vaccination with either cTIV or eTIV_a in adults and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* participation in the V58P4 study
* mentally competent to understand the nature, the scope and the consequences of the study
* able and willing to give written informed consent prior to study entry
* available for all the visits scheduled in the study

Exclusion Criteria:

* receipt of another investigational agent within 90 days prior to, or before completion of the safety follow-up period in another study, whichever is longer, prior to Visit 7 and unwilling to refuse participation in another clinical study through the end of the present study
* history of any anaphylaxis, serious vaccine reactions, or allergy to any of the vaccine components
* any acute respiratory disease or infections requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis was acceptable) or experienced fever (i.e., axillary temperature ≥ 38°C) within the 5 days prior to Visit 7
* pregnant/breast feeding women, or women of childbearing potential who refuse to use a reliable contraceptive method during the three weeks after vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1522 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (5):
- Poland (5):
  - 5, Krakow
  - 1, Krakow
  - 3, Krakow
  - 2, Krakow
  - 4, Krakow

REFERENCES:
- [Result] Szymczakiewicz-Multanowska A, Lattanzi M, Izu A, Casula D, Sparacio M, Kovacs C, Groth N. Safety assessment and immunogenicity of a cell-culture-derived influenza vaccine in adults and elderly subjects over three successive influenza seasons. Hum Vaccin Immunother. 2012 May;8(5):645-52. doi: 10.4161/hv.19493. Epub 2012 May 1. PMID 22418809
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=22418809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted during the period of October 2007 to June 2008 at five sites in Poland.
Pre-assignment Details: All subjects enrolled were included in the trial. The data entered is for overall study.
Groups:
- cTIV (Adults): Revaccination unrandomized group (adult subjects (18-60 years of age) who were pre-vaccinated in the parent (V58P4 [NCT00492063]) and the extension 1 (V58P4E1 [NCT00306527]) studies and received at least one dose of cell-culture derived seasonal trivalent influenza vaccine [cTIV] were allocated to receive cTIV or subjects who participated only in the parent study and received or were planned to receive cTIV in study E1 were allocated to receive cTIV in the deltoid muscle, preferably of the non-dominant arm).
- eTIV_a (Adults): Revaccination unrandomized group (adult subjects (18-60 years of age) who were pre-vaccinated in parent (V58P4 [NCT00492063]) and Extension 1 (V58P4E1 [NCT00306527]) studies with influenza virus vaccine[egg-derived seasonal trivalent, thiomersal free; eTIV_a] were allocated to receive eTIV_a in the deltoid muscle, preferably of the non-dominant arm).
- cTIV (Elderly): Revaccination unrandomized group (elderly subjects (>= 61 years of age) who were pre-vaccinated in parent (V58P4 [NCT00492063]) and Extension 1 (V58P4E1 [NCT00306527]) studies and received at least one dose of cell-culture derived seasonal trivalent influenza vaccine [cTIV] were allocated to receive cTIV or subjects who participated only in the parent study and received or were planned to receive cTIV in study E1 were allocated to receive cTIV in the deltoid muscle, preferably of the non-dominant arm).
- eTIV_a (Elderly): Revaccination unrandomized group (elderly subjects (>= 61 years of age) who were pre-vaccinated in parent (V58P4 [NCT00492063]) and Extension 1 (V58P4E1 [NCT00306527]) study with influenza virus vaccine [egg-derived seasonal trivalent, thiomersal free; eTIV_a] were allocated to receive eTIV_a in the deltoid muscle, preferably of the non-dominant arm).
- cTIV (Elderly; FLU Vaccination): Revaccination randomized group (elderly subjects (>= 65 years of age) were revaccinated with cell-culture derived seasonal trivalent influenza vaccine [cTIV]; in the deltoid muscle, preferably of the non-dominant arm) irrespective of influenza vaccination received in parent (V58P4 [NCT00492063]) study or extension 1 (V58P4E1 [NCT00306527]) study.
- cTIV+PV (Elderly; Concomitant Vaccination ): Revaccination randomized group (elderly subjects (>= 65 years of age) were concomitantly revaccinated with cell-culture derived seasonal trivalent influenza vaccine [cTIV; in the deltoid muscle, preferably of the non-dominant arm] and pneumococcal vaccine [PV; in opposite arm] irrespective of influenza vaccination received in parent (V58P4 [NCT00492063]) study or extension 1 (V58P4E1 [NCT00306527]) study).
- eTIV_a (Elderly; FLU Vaccination): Revaccination randomized group (elderly subjects (>= 65 years of age) were revaccinated with influenza virus vaccine [egg-derived seasonal trivalent, thiomersal free; eTIV_a] in the deltoid muscle, preferably of the non-dominant arm irrespective of influenza vaccination received in parent (V58P4 [NCT00492063]) study or extension 1 (V58P4E1 [NCT00306527]) study).
- eTIV_a +PV (Elderly; Concomitant Vaccination): Revaccination randomized group (elderly subjects (>= 65 years of age) were concomitantly revaccinated with influenza virus vaccine [egg-derived seasonal trivalent, thiomersal free; eTIV_a in the deltoid muscle, preferably of the non-dominant arm] and pneumococcal vaccine [PV; in opposite arm] irrespective of influenza vaccination received in parent (V58P4 [NCT00492063]) study or extension 1 (V58P4E1 [NCT00306527]) study).
Period: Overall Study
Arm/Group | cTIV (Adults) | eTIV_a (Adults) | cTIV (Elderly) | eTIV_a (Elderly) | cTIV (Elderly; FLU Vaccination) | cTIV+PV (Elderly; Concomitant Vaccination ) | eTIV_a (Elderly; FLU Vaccination) | eTIV_a +PV (Elderly; Concomitant Vaccination)
Started | 549 | 169 | 391 | 144 | 90 | 78 | 57 | 44
Completed | 544 | 168 | 389 | 143 | 90 | 78 | 57 | 42
Not Completed | 5 | 1 | 2 | 1 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | cTIV (Adults) | eTIV_a (Adults) | cTIV (Elderly) | eTIV_a (Elderly) | cTIV (Elderly; FLU Vaccination) | cTIV+PV (Elderly; Concomitant Vaccination ) | eTIV_a (Elderly; FLU Vaccination) | eTIV_a +PV (Elderly; Concomitant Vaccination) | Total
Number analyzed (Participants) | 549 | 169 | 391 | 144 | 90 | 78 | 57 | 44 | 1522
Age, Continuous [Mean (Standard Deviation); unit: years]
  Unrandomized adults | 44 (12.3) | 43.3 (12.4) | NA (NA) — This category does not belong to unrandomized adults | NA (NA) — This category does not belong to unrandomized adults | NA (NA) — This category does not belong to unrandomized adults | NA (NA) — This category does not belong to unrandomized adults | NA (NA) — This category does not belong to unrandomized adults | NA (NA) — This category does not belong to unrandomized adults | 43.9 (12.3)
  Unrandomized elderly | NA (NA) — This category does not belong to unrandomized elderly | NA (NA) — This category does not belong to unrandomized elderly | 71.5 (5.5) | 72.4 (5.7) | NA (NA) — This category does not belong to unrandomized elderly | NA (NA) — This category does not belong to unrandomized elderly | NA (NA) — This category does not belong to unrandomized elderly | NA (NA) — This category does not belong to unrandomized elderly | 71.7 (5.6)
  Randomized elderly | NA (NA) — This category does not belong to randomized elderly | NA (NA) — This category does not belong to randomized elderly | NA (NA) — This category does not belong to randomized elderly | NA (NA) — This category does not belong to randomized elderly | 71.6 (5.9) | 71.5 (5.5) | 71.2 (4.9) | 71.1 (5.2) | 71.4 (5.5)
Gender [Count of Participants; unit: Participants]
  Female | 318 | 102 | 232 | 90 | 46 | 40 | 38 | 25 | 891
  Male | 231 | 67 | 159 | 54 | 44 | 38 | 19 | 19 | 631

OUTCOME MEASURES:

1. Secondary Outcome: Number of Unrandomized Participants Reporting Local and Systemic Reactions.
Description: Safety and tolerability evaluation of influenza vaccines, within one week of single intramuscular injection.
Time Frame: One week postvaccination
Population: Safety set.
Measure: Number; unit: Subjects
Groups:
- cTIV (Adults): Revaccination unrandomized group (adult subjects (18-60 years of age) who were pre-vaccinated in the parent (V58P4) and the extension 1 (V58P4E1) studies and received at least one dose of cell-culture derived seasonal trivalent influenza vaccine (cTIV) were allocated to receive cTIV or subjects who participated only in the parent study and received or were planned to receive cTIV in study E1 were allocated to receive cTIV in the deltoid muscle, preferably of the non-dominant arm).
- eTIV_a (Adults): Revaccination unrandomized group (adult subjects (18-60 years of age) who were pre-vaccinated in parent (V58P4) and Extension 1 (V58P4E1) studies with influenza virus vaccine(egg-derived seasonal trivalent, thiomersal free; eTIV_a) were allocated to receive eTIV_a in the deltoid muscle, preferably of the non-dominant arm).
- cTIV (Elderly): Revaccination unrandomized group (elderly (>= 61 years of age)subjects who were pre-vaccinated in parent (V58P4) and Extension 1 (V58P4E1) studies and received at least one dose of cell-culture derived seasonal trivalent influenza vaccine (cTIV) were allocated to receive cTIV or subjects who participated only in the parent study and received or were planned to receive cTIV in study E1 were allocated to receive cTIV in the deltoid muscle, preferably of the non-dominant arm).
- eTIV_a (Elderly): Revaccination unrandomized group (elderly (>= 61 years of age)subjects who were pre-vaccinated in parent (V58P4) and Extension 1 (V58P4E1) study with influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a) were allocated to receive eTIV_a in the deltoid muscle, preferably of the non-dominant arm).
Arm/Group | cTIV (Adults) | eTIV_a (Adults) | cTIV (Elderly) | eTIV_a (Elderly)
Number analyzed (Participants) | 550 | 168 | 391 | 144
Subjects
  Local Reactions | 185 | 60 | 98 | 26
  Erythema | 50 | 20 | 36 | 10
  Induration | 38 | 14 | 26 | 3
  Swelling | 23 | 7 | 17 | 3
  Ecchymosis | 12 | 1 | 14 | 2
  Pain | 158 | 51 | 64 | 12
  Systemic Reaction | 99 | 28 | 57 | 25
  Chills | 15 | 5 | 5 | 4
  Malaise | 52 | 16 | 37 | 16
  Myalgia | 40 | 8 | 25 | 8
  Arthralgia | 18 | 5 | 16 | 6
  Headache | 39 | 18 | 20 | 11
  Sweating | 18 | 8 | 13 | 8
  Fatigue | 35 | 11 | 23 | 11
  Fever (≥ 38°C) | 2 | 2 | 0 | 0
  Analgesic and Antipyretics used | 17 | 11 | 7 | 6
  Stay at Home Due to Vaccination Reaction | 5 | 5 | 6 | 3

2. Secondary Outcome: Number of Randomized Participants Reporting Local and Systemic Reactions.
Description: Safety and tolerability evaluation, within one week of single intramuscular injection of influenza vaccines (cell-culture derived seasonal trivalent influenza vaccine (cTIV) or influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a) when administered alone or concomitantly with a pneumococcal vaccine (PV)). Local reactions reported for Influenza Vaccine Injection Site.
Time Frame: One week postvaccination
Description (as registered): Safety and tolerability evaluation of influenza vaccines, within one week of single intramuscular injection. Local reactions reported for Influenza Vaccine Injection site.
Population: Safety Set
Measure: Number; unit: Subjects
Groups:
- FLU (cTIV or eTIV_a) + PV: Elderly subjects (>= 65 years of age) randomized and received influenza vaccine (cell-culture derived seasonal trivalent influenza vaccine (cTIV) or influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a) concomitantly with pneumococcal vaccine (PV)).
- FLU (cTIV or eTIV_a): Elderly subjects (>= 65 years of age) randomized and received only Influenza vaccine (cell-culture derived seasonal trivalent influenza vaccine (cTIV) or influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a)).
- cTIV (Elderly; FLU Vaccination): Revaccination randomized group (elderly subjects (>= 65 years of age) were revaccinated with cell-culture derived seasonal trivalent influenza vaccine (cTIV; in the deltoid muscle, preferably of the non-dominant arm) irrespective of influenza vaccination received in parent (V58P4) study or extension 1 (V58P4E1) study.
- cTIV+PV (Elderly; Concomitant Vaccination ): Revaccination randomized group (elderly subjects (>= 65 years of age) were concomitantly revaccinated with cell-culture derived seasonal trivalent influenza vaccine (cTIV; in the deltoid muscle, preferably of the non-dominant arm) and pneumococcal vaccine (PV; in opposite arm) irrespective of influenza vaccination received in parent (V58P4) study or extension 1 (V58P4E1) study).
- eTIV_a (Elderly; FLU Vaccination): Revaccination randomized group (elderly subjects (>= 65 years of age) were revaccinated with influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a) in the deltoid muscle, preferably of the non-dominant arm irrespective of influenza vaccination received in parent (V58P4) study or extension 1 (V58P4E1) study).
- eTIV_a+PV (Elderly; Concomitant Vaccination): Revaccination randomized group (elderly subjects (>= 65 years of age) were concomitantly revaccinated with influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a) in the deltoid muscle, preferably of the non-dominant arm) and pneumococcal vaccine (PV; in opposite arm) irrespective of influenza vaccination received in parent (V58P4) study or extension 1 (V58P4E1) study).
Arm/Group | FLU (cTIV or eTIV_a) + PV | FLU (cTIV or eTIV_a) | cTIV (Elderly; FLU Vaccination) | cTIV+PV (Elderly; Concomitant Vaccination ) | eTIV_a (Elderly; FLU Vaccination) | eTIV_a+PV (Elderly; Concomitant Vaccination)
Number analyzed (Participants) | 134 | 135 | 83 | 84 | 52 | 50
Subjects
  Local Reactions | 49 | 40 | 20 | 32 | 20 | 17
  Ecchymosis | 7 | 8 | 3 | 3 | 5 | 4
  Erythema | 20 | 23 | 12 | 12 | 11 | 8
  Induration | 9 | 14 | 9 | 6 | 5 | 3
  Swelling | 6 | 10 | 6 | 3 | 4 | 3
  Pain | 31 | 19 | 11 | 23 | 8 | 8
  Systemic Reaction | 29 | 19 | 10 | 22 | 9 | 7
  Chills | 6 | 5 | 2 | 3 | 3 | 3
  Malaise | 19 | 9 | 6 | 14 | 3 | 5
  Myalgia | 8 | 9 | 6 | 8 | 3 | 0
  Arthralgia | 14 | 9 | 6 | 11 | 3 | 3
  Headache | 12 | 9 | 4 | 11 | 5 | 1
  Sweating | 6 | 7 | 4 | 5 | 3 | 1
  Fatigue | 10 | 7 | 6 | 10 | 1 | 0
  Fever (≥ 38°C) | 0 | 0 | 0 | 0 | 0 | 0
  Analgesic and Antipyretics used | 8 | 8 | 5 | 6 | 3 | 2
  Stayed at Home Due to Vaccination Reaction | 2 | 0 | 0 | 2 | 0 | 0

3. Primary Outcome: Number of Randomized Participants Reporting Local and Systemic Reactions.
Description: Safety and tolerability evaluation of influenza vaccines, within one week of single intramuscular injection. Local reactions reported for Influenza Vaccine Injection site.
Time Frame: One week postvaccination
Description (as registered): Safety and tolerability evaluation, within one week of single intramuscular injection of influenza vaccines (cell-culture derived seasonal trivalent influenza vaccine (cTIV) or influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a) when administered alone or concomitantly with a pneumococcal vaccine (PV)). Local reactions reported for Influenza Vaccine Injection Site.
Population: Safety set: this population consisted of all subjects who were vaccinated and who had some post-baseline safety data.
Measure: Number; unit: Subjects
Groups:
- cTIV Total (Elderly): Revaccination randomized group total (elderly subjects (>= 65 years of age) who received only cell-culture derived seasonal trivalent influenza vaccine (cTIV) in the deltoid muscle, preferably of the non-dominant arm; or received concomitant pneumococcal vaccine (PV; in opposite arm)).
- eTIV_a Total (Elderly): Revaccination randomized group total (elderly subjects (>= 65 years of age) who received only influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a) in the deltoid muscle, preferably of the non-dominant arm; or received concomitant pneumococcal vaccine (PV; in opposite arm)).
Arm/Group | cTIV Total (Elderly) | eTIV_a Total (Elderly)
Number analyzed (Participants) | 167 | 102
Subjects
  Local Reactions | 52 | 37
  Erythema | 24 | 19
  Induration | 15 | 8
  Swelling | 9 | 7
  Ecchymosis | 6 | 9
  Pain | 34 | 16
  Systemic Reaction | 32 | 16
  Chills | 5 | 6
  Malaise | 20 | 8
  Myalgia | 14 | 3
  Arthralgia | 17 | 6
  Headache | 15 | 6
  Sweating | 9 | 4
  Fatigue | 16 | 1
  Fever (≥ 38°C) | 0 | 0
  Analgesic and Antipyretics used | 11 | 5
  Stayed at Home Due to Vaccination Reaction | 2 | 0

4. Secondary Outcome: Number of Subjects With Antibody Response as Assessed by Hemagglutination Inhibition Assay.
Description: Immunogenicity (seroconversion or significant increase in antibody titer and HI titer ≥1:40) of cell cultured and egg based trivalent influenza vaccine three weeks after a single injection, by the measurement of strain-specific hemagglutination inhibition (HI) tests according to the Committee for Medicinal Products for Human Use (CHMP) criteria (CPMP/BWP/214/96).
  Seroconversion was defined as negative pre-vaccination titer (<10)/postvaccination titer ≥40. Significant increase in antibody titer was defined as at least a fourfold increase from non-negative baseline (≥10).
Time Frame: Three weeks postvaccination
Population: Per Protocol Set
Measure: Number; unit: Subjects
Groups:
- cTIV (Adults): Revaccination unrandomized group (adult subjects (18-60 years of age) who were pre-vaccinated in the parent (V58P4 [NCT00492063]) and the extension 1 (V58P4E1 [NCT00306527]) studies and received at least one dose of cell-culture derived seasonal trivalent influenza vaccine (cTIV) were allocated to receive cTIV or subjects who participated only in the parent study and received or were planned to receive cTIV in study E1 were allocated to receive cTIV in the deltoid muscle, preferably of the non-dominant arm).
- eTIV_a (Adults): Revaccination unrandomized group (adult subjects (18-60 years of age) who were pre-vaccinated in parent (V58P4 [NCT00492063]) and Extension 1 (V58P4E1 [NCT00306527]) studies with influenza virus vaccine(egg-derived seasonal trivalent, thiomersal free; eTIV_a) were allocated to receive eTIV_a in the deltoid muscle, preferably of the non-dominant arm).
- cTIV Total (Elderly): Revaccination randomized group total (elderly subjects (>= 61 years of age) who received only (cell-culture derived seasonal trivalent influenza vaccine (cTIV) in the deltoid muscle, preferably of the non-dominant arm; or received concomitant pneumococcal vaccine (PV; in opposite arm)).
- eTIV_a Total (Elderly): Revaccination randomized group total (elderly subjects (>= 61 years of age) who received only influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a) in the deltoid muscle, preferably of the non-dominant arm; or received concomitant pneumococcal vaccine (PV; in opposite arm)).
Arm/Group | cTIV (Adults) | eTIV_a (Adults) | cTIV Total (Elderly) | eTIV_a Total (Elderly)
Number analyzed (Participants) | 95 | 23 | 89 | 62
Subjects
  HI titer ≥1:40 (H1N1) | 94 | 23 | 85 | 55
  seroconversion (H1N1) | 57 | 13 | 62 | 41
  HI titer ≥1:40 (H3N2) | 92 | 22 | 86 | 59
  seroconversion (H3N2) | 40 | 8 | 32 | 25
  HI titer ≥1:40 (B) | 57 | 16 | 56 | 33
  seroconversion (B) | 39 | 8 | 23 | 18

5. Secondary Outcome: Geometric Mean Ratio (GMR Day 22/Day1) After Single Dose of Influenza Vaccine.
Description: Immunogenicity (geometric mean titer ratio) of cell cultured and egg based trivalent influenza vaccine three weeks after a single injection, by the measurement of strain-specific hemagglutination inhibition (HI) tests according to the CHMP criteria (CPMP/BWP/214/96).
  CHMP Criteria fulfilled if the Geometric Mean titer Ratio (GMR) is > 2.5.
Time Frame: Three weeks postvaccination
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | cTIV (Adults) | eTIV_a (Adults) | cTIV Total (Elderly) | eTIV_a Total (Elderly)
Number analyzed (Participants) | 95 | 23 | 89 | 62
Ratio
  GMR (H1N1; A/Solomon Islands/3/2006) | 5.6 [4.27 to 7.34] | 4.38 [2.52 to 7.6] | 7.75 [5.93 to 10] | 5.92 [4.29 to 8.16]
  GMR (H3N2; A/Wisconsin/67/2005) | 3.63 [2.83 to 4.64] | 2.33 [1.41 to 3.85] | 2.65 [2.22 to 3.16] | 2.89 [2.34 to 3.58]
  GMR (B; B/Malaysia/2506/2004) | 4.48 [3.43 to 5.84] | 2.33 [1.35 to 3.99] | 2.51 [1.96 to 3.21] | 2.97 [2.21 to 4]

6. Primary Outcome: Immunogenicity Assessment by Geometric Mean Titers (GMT).
Description: Non-inferiority of the influenza vaccine FLU (cell-culture derived seasonal trivalent influenza vaccine (cTIV); and influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a)) when administered alone versus administered concomitantly with pneumococcal vaccine (FLU + PV) is met if lower limit of the 2-sided 95% confidence interval (CI) of postvaccination (Day 22) Geometric Mean Titer ratio (FLU+PV/FLU) is greater than 0.5.
Time Frame: Three weeks postvaccination
Population: Per protocol set: this population consisted of all subjects in the Intention To Treat population (ITT) who had no major protocol violation as defined prior to analysis (ITT=enrolled subjects who received single dose of influenza vaccine(or 2 vaccines if receiving the pneumococcal vaccine) and provided one serum sample before and one after baseline)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- FLU (cTIV or eTIV_a) + PV: Elderly subjects (>= 65 years of age) randomized and received influenza vaccine (cell-culture derived seasonal trivalent influenza vaccine (cTIV) or influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a) concomitantly with pneumococcal vaccine (PV).
- FLU (cTIV or eTIV_a): Elderly subjects (>= 65 years of age) randomized and received only Influenza vaccine (cell-culture derived seasonal trivalent influenza vaccine (cTIV) or influenza virus vaccine (egg-derived seasonal trivalent, thiomersal free; eTIV_a).
Arm/Group | FLU (cTIV or eTIV_a) + PV | FLU (cTIV or eTIV_a)
Number analyzed (Participants) | 74 | 77
Titers
  GMT Day 22 (H1N1) | 138 [104 to 182] | 198 [151 to 259]
  GMT Day 22 (H3N2) | 184 [141 to 240] | 228 [176 to 296]
  GMT Day 22 (B) | 36 [27 to 47] | 52 [40 to 68]
Statistical Analysis 1: Comparison: FLU (cTIV or eTIV_a) + PV vs FLU (cTIV or eTIV_a); The non-inferiority null hypothesis stated that the FLU+PV vaccine group was non-inferior to the FLU alone group if the lower limit of the 95% CI of the ratio of GMTs between vaccines (FLU+PV/FLU alone) on day 22 was greater than 0.5 for all three vaccine strains; Test type: Non-Inferiority or Equivalence — Non-inferiority was met if lower limit of the 2-sided 95% Clopper-Pearson confidence interval (CI) of the ratio of the postvaccination (Day 22) Geometric Mean Titers (FLU+PV/FLU vaccine alone) was greater than 0.5; Ratio of GMTs = 0.66, 95% CI 2-sided [0.45 to 0.98] — A/H1N1(Day22)
Statistical Analysis 2: Comparison: FLU (cTIV or eTIV_a) + PV vs FLU (cTIV or eTIV_a); [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio of GMTs = 0.81, 95% CI 2-sided [0.55 to 1.19] — A/H3N2 (Day 22)-criterion was met
Statistical Analysis 3: Comparison: FLU (cTIV or eTIV_a) + PV vs FLU (cTIV or eTIV_a); [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio of GMTs = 0.69, 95% CI 2-sided [0.46 to 1.02] — B (Day 22)

ADVERSE EVENTS:
Time Frame: Throughout the entire study period (six months)
Description: Other Adverse Events (AEs) (>5%) includes solicited local and systemic reactions collected within the first 7 days following vaccination along with unsolicited AEs collected within first three weeks after the vaccination. Local reactions for groups cTIV+PV and eTIV_a+PV were collected for influenza vaccine and pneumococcal vaccine injection sites.
Groups:
- cTIV+PV (Elderly; Concomitant Vaccination ): Revaccination randomized group (elderly subjects (>= 65 years of age)were concomitantly revaccinated with cell-culture derived seasonal trivalent influenza vaccine [cTIV; in the deltoid muscle, preferably of the non-dominant arm] and pneumococcal vaccine [PV; in opposite arm] irrespective of influenza vaccination received in parent (V58P4 [NCT00492063]) study or extension 1 (V58P4E1 [NCT00306527]) study).
- eTIV_a (Elderly; FLU Vaccination): Revaccination randomized group (elderly subjects (>= 65 years of age)were revaccinated with influenza virus vaccine [egg-derived seasonal trivalent, thiomersal free; eTIV_a] in the deltoid muscle, preferably of the non-dominant arm irrespective of influenza vaccination received in parent (V58P4 [NCT00492063]) study or extension 1 (V58P4E1 [NCT00306527]) study).
Arm/Group | cTIV (Adults) | eTIV_a (Adults) | cTIV (Elderly) | eTIV_a (Elderly) | cTIV (Elderly; FLU Vaccination) | cTIV+PV (Elderly; Concomitant Vaccination ) | eTIV_a (Elderly; FLU Vaccination) | eTIV_a +PV (Elderly; Concomitant Vaccination)
Serious Adverse Events (participants affected / at risk) | 17/550 | 5/168 | 23/391 | 6/144 | 3/83 | 5/84 | 1/52 | 6/50
Other Adverse Events (participants affected / at risk) | 219/550 | 73/168 | 119/391 | 40/144 | 25/83 | 48/84 | 23/52 | 21/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | cTIV (Adults) (N=550) | eTIV_a (Adults) (N=168) | cTIV (Elderly) (N=391) | eTIV_a (Elderly) (N=144) | cTIV (Elderly; FLU Vaccination) (N=83) | cTIV+PV (Elderly; Concomitant Vaccination ) (N=84) | eTIV_a (Elderly; FLU Vaccination) (N=52) | eTIV_a +PV (Elderly; Concomitant Vaccination) (N=50)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infraction (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infraction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inner ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iridocele (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitreous prolapse (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diagnostic procedure (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurilemmoma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Motor neurone disease (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arteriosclerosis obliterans (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervix adenomatous polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | cTIV (Adults) (N=550) | eTIV_a (Adults) (N=168) | cTIV (Elderly) (N=391) | eTIV_a (Elderly) (N=144) | cTIV (Elderly; FLU Vaccination) (N=83) | cTIV+PV (Elderly; Concomitant Vaccination ) (N=84) | eTIV_a (Elderly; FLU Vaccination) (N=52) | eTIV_a +PV (Elderly; Concomitant Vaccination) (N=50)
Chills (General disorders) | 15 | 5 | 5 | 4 | 2 | 3 | 3 | 3
Fatigue (General disorders) | 35 | 11 | 23 | 11 | 7 | 10 | 2 | 0
Injection site erythema (General disorders) | 50 | 20 | 36 | 10 | 12 | 19 | 11 | 8
Injection site haemorrhage (General disorders) | 12 | 1 | 14 | 2 | 3 | 5 | 5 | 5
Injection site induration (General disorders) | 38 | 14 | 26 | 3 | 9 | 11 | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 5 | 16 | 6 | 7 | 11 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 41 | 8 | 25 | 8 | 6 | 8 | 3 | 0
Headache (Nervous system disorders) | 42 | 19 | 20 | 11 | 5 | 12 | 5 | 1
Injection site swelling (General disorders) | 23 | 7 | 17 | 3 | 6 | 4 | 4 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 18 | 8 | 13 | 8 | 5 | 5 | 3 | 1
Injection site pain (General disorders) | 158 | 51 | 64 | 12 | 11 | 32 | 8 | 10
Malaise (General disorders) | 52 | 16 | 37 | 16 | 7 | 14 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days